CLINICAL TRIAL: NCT00240877
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of a Monovalent Vaccine of a New 6:2 Reassortant in Healthy Adults (AV024)
Brief Title: Study to Evaluate the Safety of a Monovalent Vaccine of a New 6:2 Reassortant in Healthy Adults (AV024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Robert Walker, M.D., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AV024
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Monovalent vaccine prior to the release of the trivalent vaccine (FluMist).
  Interventions: Biological: AV024
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AV024 — 0.5 mL total dose volume administered intranasal by spray applicator (approximately 0.25 mL into each nostril).
  Arms: 1
Other: Placebo — Placebo mist consisting of normal allantoic fluid. 0.5 mL total dose volume administered intranasal by spray applicator (approximately 0.25 mL into each nostril).
  Arms: 2

SUMMARY:
To assess the safety of a vaccine in healthy adults prior to the release of the trivalent vaccine (FluMist).

DETAILED DESCRIPTION:
The primary study objective is to assess the safety of a monovalent vaccine of a new 6:2 reassortant in healthy adults prior to the release of the trivalent vaccine (FluMist). Safety will be demonstrated by similar fever rates (oral temperature ≥101°F) in vaccine and placebo recipients.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age (not yet reached their 65th birthday);
* In good health;
* Available by telephone;
* Ability to understand and comply with the requirements of the protocol; and
* Signed informed consent.

Exclusion Criteria:

* Any condition, other than age, for which the inactivated influenza vaccine is indicated, including: chronic disorders of the pulmonary or cardiovascular systems, including asthma; chronic metabolic diseases (including diabetes mellitus) renal dysfunction, or hemoglobinopathies which required regular medical follow-up or hospitalization during the proceeding year;
* Acute febrile (>100.0°F oral) illness or clinically significant respiratory illness within the 14 days prior to enrollment;
* Hypersensitivity to egg or egg protein;
* Signs or symptoms of any immunosuppressive or immune deficiency disease, including HIV infection, or ongoing immunosuppressive therapy; or an immunosuppressed individual living in the same household;
* Participation in another investigational trial within one month prior to enrollment or expected enrollment in another investigational trial during this study; and
* Any condition that in the opinion of the investigator, might interfere with the vaccine evaluation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2002-08; Primary Completion 2003-08 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
- The primary endpoint of this study is fever defined as oral temperature ≥101°F | Days 0-7

SECONDARY OUTCOMES:
All other reported reactogenicity events and other adverse events. | After 7 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- SFBC International Inc, Miami, Florida, United States